CLINICAL TRIAL: NCT05772104
Title: A Multi-center, Randomized, Double-Blind Clinical Trial of Shugan Jieyu Capsule in Generalized Anxiety Disorder
Brief Title: Clinical Trial of Shugan Jieyu Capsule in Generalized Anxiety Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Jishengtang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH109-CS01-CRP
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Shugan Jieyu Capsules (Experimental): Participants received Shugan Jieyu Capsules 4 capsules,BID,once in the morning and once in the evening, at an interval of more than 8 hours, for up tp 12 weeks.
  Interventions: Drug: Shugan Jieyu Capsules
- Experimental: Shugan Jieyu Capsules Placepo (Placebo Comparator): Participants received Shugan Jieyu Capsules Placebo 4 capsules,BID,once in the morning and once in the evening, at an interval of more than 8 hours, for up tp 12 weeks.
  Interventions: Drug: Shugan Jieyu Capsules Placebo

INTERVENTIONS:
Drug: Shugan Jieyu Capsules — Oral, 4 Capsules, BID
  Arms: Experimental: Shugan Jieyu Capsules
Drug: Shugan Jieyu Capsules Placebo — Drug: Shugan Jieyu Capsules Placebo, Oral，4 capsules，BID
  Drug: Placebo, Oral, 1 capsule, BID
  Arms: Experimental: Shugan Jieyu Capsules Placepo

SUMMARY:
This is a randomized double-blind placebo-controlled phase 3 clinical trial to further validate the effectiveness and safety of Shugan Jieyu Capsules in treating generalized anxiety disorder.

DETAILED DESCRIPTION:
This trial was a multi-center, randomized, double-blind, two-stage clinical trial in patients with generalized anxiety disorder (TCM differentiated as liver Qi stagnation and spleen deficiency syndrome), consisting of a exploratory study(stage 1) and a confirmatory study(stage 2).

In stage 1, 120 subjects were enrolled and randomly assigned to high-dose group, low-dose group and placebo group at a ratio of 1:1:1.

In stage 2, 495 subjects were randomly assigned to the experimental and placebo groups at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of generalized anxiety disorder (GAD) as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) as confirmed by the MINI at Screening, The duration of illness must be ≥ 6 months；
2. Age 18-65 years old；
3. Hamilton Anxiety Rating Scale (HAM-A) Total Score of ≥ 14 at both Screening and Baseline，Anxious Mood (item 1) score ≥2；
4. Clinical Global Impression of Severity Scale (CGI-S) score of ≥ 3 at both Screening and Baseline
5. The TCM syndrome is liver Qi stagnation and spleen deficiency syndrome.

Exclusion Criteria:

1. Diagnosed with a psychiatric disorder other than GAD that meets DSM-5 criteria within 6 months prior to screening；
2. Alcohol or drug abuse or dependence in the 6 months prior to screening, or urine positive for multiple drugs combined at screening
3. Hamilton Depression Rating Scale (HAMD-17) Total Score of > 17 at Screening or Baseline，or Depressive Mood (item 1) score ≥2；
4. Patients with Severe Insomnia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the HAM-A Total Score at Week 12 | Change from Baseline to Week 12
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.

SECONDARY OUTCOMES:
Change From Baseline in the HAM-A Total Score at Week 2, 4, and 8 | Change from Baseline to Week 2, 4, and 8
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
The Proportion of Subjects with HAM-A Total Score Reduction Rate ≥50% at week 2, 4, 8 and 12; | Change from Baseline to Week 2, 4, 8 and 12
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
The Proportion of Subjects with HAM-A Total Score ≤7 at week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
Change From Baseline in the HAM-A Mental Anxiety Score at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  HAM-A Mental Anxiety Score was the sum of Items 1 to 6 and Item 14 and could have ranged from 0 to 28.
Change From Baseline in the HAM-A Somatic Anxiety Score at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  The HAM-A Somatic Anxiety Factor Score was the sum of Items 7 to 13 and could have ranged from 0 to 28.
Change From Baseline in the The World Health Organization Quality of Life (WHOQOL)-BREF at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  The scale evaluates the quality of life in four areas: physiology, psychology, social relations and environment.
Change From Baseline in the Clinical Global Impression of Severity Scale (CGI-S) at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  The CGI-S is measures the clinician's impression of a subject's current anxiety severity considering their total clinical experience with the patient population. This measure uses a 0-7 scale, with higher scores indicating greater anxiety severity.
Change From Baseline in the Clinical Global Impression of Improvement Scale (CGI-I) at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  CGI-I measured the clinician's perception of the participant's improvement at the time of assessment compared with the baseline. Scores could have ranged from 1 (very much improved) to 7 (very much worse).
Change From Baseline in the Traditional Chinese Medicine Syndrome Score Scale at Week 2, 4, 8 and 12 | Change from Baseline to Week 2, 4, 8 and 12
  TCM syndrome scale was used to evaluate the changes of TCM symptoms and signs before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD, Principal Investigator — Beijing Anding Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No